CLINICAL TRIAL: NCT05530603
Title: Intervention to Promote Breast Cancer Screening Among American Indian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Collaborators: University of North Dakota (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Soonhee Roh, Professor, University of South Dakota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-053; U54GM128729 (NIH)
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 arms randomized clinical trial with control and intervention group
Who Masked: Participant
Masking Description: Participants are unaware of which group they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants are randomized to interventional arm which is seven-day intervention that requires them to download mobile app to complete educational courses each day. Participants are required to complete pre- and post-tests as part of the study. The intervention encourages education on mammogram needs.
  Interventions: Behavioral: Educational mobile app
- Control (No Intervention): Participants are randomized to control arm where they are give an education brochure. There are pre and post tests to complete.

INTERVENTIONS:
Behavioral: Educational mobile app — 7 day educational course to educate American Indian women to receive regular mammogram.
  Arms: Intervention

SUMMARY:
Our objectives in this project are to develop and evaluate the feasibility and effectiveness of the Mobile Web App Breast Cancer Screening (wMammogram) intervention that is culturally tailored for AI women residing in rural areas. The proposed study will be a multi-method, two-phase research project that will take place in South Dakota over a three-year period. The two phases are: (1) developing the wMammogram intervention and (2) evaluating the feasibility and efficacy of the wMammogram. Phase 1 incorporates a community-based participatory research approach and a series of focus groups with various stakeholders in American Indian (AI) communities to design a culturally informed and practically refined intervention. Phase 2 uses a randomized clinical trial (RCT) design with AI women. The wMammogram intervention will be applied throughout a seven-day period, with assessment at three intervals: baseline (survey), one-week post-intervention (survey), and six-month follow-up (telephone survey).

The wMammogram intervention will be implemented with AI women using the two-arm RCT that includes recruiting a total of 120 AI women aged 40 to 70 years and randomly assigning them to either (a) the wMammogram intervention group (n=60) to receive culturally and personally tailored multilevel and multimedia messages through a Mobile Web App along with health navigator services or (b) the control group (n=60) to receive the mailing of printed educational materials on breast cancer and relevant screening guidelines along with health navigator services.

Hypotheses: In assessing the efficacy and feasibility of the wMammogram, Investigators hypothesize that:

(H1)The wMammogram intervention participants will show a higher rate of mammograms received than will participants in the educational materials intervention.

(H2)The wMammogram intervention participants will show improvements in knowledge, attitude, and beliefs about breast cancer screening and readiness for mammography as compared to participants in the educational materials intervention.

(H3)The wMammogram intervention participants will demonstrate greater satisfaction with and acceptance of the intervention than would participants in the educational materials intervention.

DETAILED DESCRIPTION:
Sample Size and Power Analysis: Investigators will have 120 participants in both the intervention and the control group by the six-month follow-up assessment. Considering that the possible sample attrition at the six-month follow-up is expected to be no higher than 20% (n=24), a total of 144 participants will be recruited for the baseline assessment; half will be randomly assigned to intervention (n=72) and another half assigned to control condition (n=72). Using a one-sided nonparametric Wilcoxon rank-sum test and the mixed effect ANOVA at the 0.05 level and assuming continuous scores, this sample size (60 per arm) would provide 80 percent power to reject the null hypothesis of the equality of score-changes for both groups. The key objective of the study is to acquire preliminary estimates of breast cancer screening rates after the intervention to assess if further study is warranted. As such, Investigators stress on the precision with which Investigators can estimate the breast cancer screening rate post-intervention rather than our ability to reject a specific null hypothesis. A sample size of 60 participants for each arm reflects a compromise between keeping the scope of the project within the objectives of a pilot study while ensuring a large enough sample size to estimate the breast cancer screening rate post-intervention.

Quantitative Measures (Baseline, One-Week, and Six-Month Follow-Up Assessment): Measures will be selected based on the frequency of use in cancer and health literature, psychometric properties, previous applications with AI populations, and inputs from the Community Advisory Board (CAB) and focus groups. The primary outcome criterion for efficacy is mammography receipt after the intervention, which will be measured by self-report (yes or no) at six-month follow-up. The measure has been widely used and found reliable in cancer screening research. The secondary outcome criteria for efficacy include breast cancer knowledge, health beliefs, cultural attitudes, and intent to undergo screening. These measures will be administered at multiple points: baseline and one-week post-intervention. In order to assess feasibility, investigators will measure participant satisfaction and intervention effectiveness. These measures will be administered at one week after the intervention. Confounding covariates (e.g., background, sociodemographic, and health-related information) will be collected only at the baseline assessment and used for assessing the influence of such contextual factors.

Quantitative Data Analysis: Prior to our hypotheses tests, group equivalence in terms of baseline characteristics will be examined using t-tests and chi-square tests. For Hypothesis 1, Investigators will compare the percentage of women from each condition who receive mammograms or have scheduled a mammography appointment using a chi-square test. Investigators will supplement this with logistic regression analyses to adjust for confounding covariates. For Hypothesis 2, the averages of score change (pre- to post-test) from the two conditions will be compared using the two-sample t-test, and/or the Wilcoxon rank-sum tests after assessing normality of the scores. The group difference in terms of changes in the given constructs will be tested by a mixed-effect analysis of variance (ANOVA). The mixed-effect ANOVA includes both within-subject (i.e., time: repeated measures) and between-subject factors (i.e., group: intervention versus control) and aims to examine whether there is an interaction between these two factors on the dependent variable. Bonferroni correction will be used to reduce the probability of Type 1 error for multiple comparisons. Investigators will supplement this with a regression analysis of score change in order to adjust for confounding covariates. For Hypothesis 3, averages of general satisfaction and effectiveness scores from each group will be compared using the two-sample t-test. Also, the percentage of participants from each group who endorse "yes" for the intention and recommendation items will be compared using the chi-square test. To minimize a potential non-participation bias, Investigators will closely monitor and compare the first and fourth quartiles of responses for differences in background variables and key constructs. Investigators will also carefully document the response rate over the course of this project. IBM SPSS version 25 will be used for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women who are self-identified AI women of the YST in SD
* Women who are aged 40 to 70 years
* Women who have not received a mammogram in the past two years
* Women who are willing to use their own mobile phone, iPad, tablets, and computers, or a mobile phone borrowed from the research team for the wMammogram intervention.

Exclusion Criteria:

* Women who received a mammogram in the past year
* Women who are under 40 or over 70 years of age.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-10-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SOONHEE ROH, PhD, Principal Investigator — University of South Dakota
Locations (2):
- United States (2):
  - Yankton Sioux Tribe, Lake Andes, South Dakota
  - University of South Dakota, Vermillion, South Dakota

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD with other researchers

REFERENCES:
- [Derived] Roh S, Lee YS, Kenyon DB, Elliott AJ, Petereit DG, Gaba A, Lee HY. Mobile Web App Intervention to Promote Breast Cancer Screening Among American Indian Women in the Northern Plains: Feasibility and Efficacy Study. JMIR Form Res. 2023 Jul 20;7:e47851. doi: 10.2196/47851. PMID 37471115

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 66 | 67
Completed | 62 | 60
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 66 | 67 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 56 | 115
  >=65 years | 7 | 11 | 18
Age, Continuous [Mean (Full Range); unit: years] | 50.50 [40 to 70] | 55.37 [40 to 70] | 52.89 [40 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 67 | 133
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 66 | 67 | 133
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 67 | 133
Receipt of Mammogram [Count of Participants; unit: Participants] | 26 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received a Mammogram
Description: This outcome was assessed based on the number of participants who reported having received a mammogram during the six-month follow-up survey. The survey asked participants, "Have you ever received a mammogram since you had participated in a mammogram intervention?" Participants could respond with either "Yes, I have received one" or "No, I haven't received one yet." We calculated and compared the number of participants from each arm who received mammograms after the intervention.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
Participants | 26 | 12
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .009, Chi-squared — The threshold for statistical significance was p=0.05

2. Secondary Outcome: Change in Participants' Breast Cancer Knowledge Levels From Baseline to Week 1
Description: Participants' breast cancer knowledge levels were assessed using the Breast Cancer Knowledge Test, which includes 28 true- or false-items. Scores were determined by the number of correct responses, with the total score ranging from 0 to 28. Higher scores indicate greater breast cancer knowledge, with a score of 0 reflecting no knowledge and a score of 28 indicating very high knowledge. The test was updated to align with the latest American Cancer Society breast cancer screening guideline. Change = (Week 1 Score - Baseline Score).
Time Frame: Baseline and Week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
units on a scale | 22.95 (4.58) | 21.83 (4.52)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = 0.730, ANOVA — The threshold for statistical significance was p=0.05; Mean Difference (Net) = 1.12, Standard Deviation 0.80

3. Secondary Outcome: Health Beliefs
Description: Participants' health beliefs were assessed using a 5-item prevention orientation scale at one week post-intervention. The scale included items, such as "Even if I do not have a family history of cancer, it is important to be checked regularly," and "It is better to detect health problems early through screening efforts than discover something later and have to treat it." Each item was rated on a 4-point Likert scale, ranging from "1=strongly disagree" to "4=strongly agree." Scores for each item were calculated by summing the item responses, with total scores ranging from 5 to 20. Higher item scores indicated stronger health beliefs related to prevention orientation. Change = (Week 1 Score - Baseline Score).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
units on a scale | 10.19 (1.678) | 9.95 (1.692)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .033, ANOVA — The threshold for statistical significance was p=0.05

4. Secondary Outcome: Cultural Attitudes
Description: Cultural attitudes toward breast cancer screening were assessed using a 6-items cultural modesty scale. Each item was rated on a 4-point scale, ranging from "1=strongly disagree" to "4=strongly agree." Higher item scores indicated stronger belief in cultural modesty. The total score for each item was computed by summing the individual item scores, ranging from 6 to 24.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
units on a scale | 11.85 (3.067) | 12.60 (3.509)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .068, ANOVA; The threshold for statistical significance was p=0.05

5. Secondary Outcome: Number of Participants Who Intended to Receive a Mammogram in the Future
Description: Number of Participants who intended to receive a mammogram in the future was assessed by a single question at both baseline and 1 week after the intervention. The single question asked whether a participant intended to receive a mammogram in the future, with response options of "0=No intention" or "1=Yes intention." The data values represent the number of participants who intended to receive a mammogram in the future with the response of "Yes intention."
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
Participants | 62 | 51
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .001, Fisher Exact — The threshold for statistical significance was p=0.05

6. Secondary Outcome: Number of Participants Satisfied With Intervention
Description: Number of participants satisfied with intervention they received was assessed using a 2-point scale ranging from "1=Dissatisfied/Very dissatisfied" to "2=Satisfied/Very Satisfied" one week after the intervention. The data values represent the number of participants satisfied with intervention with response option of "2=Satisfied/Very Satisfied."
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
Participants | 60 | 53
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .001, t-test, 2 sided — The threshold for statistical significance was p=0.05

7. Secondary Outcome: Number of Participants Indicating Intervention Was Effective/Very Effective
Description: Number of Participants Indicating Intervention Was Effective/Very Effective was measured one week after the intervention with the question, "Do you think that the intervention you received was effective in increasing your knowledge of breast cancer and screenings?" Participants responded on a 4-point scale item ranging from "1=very ineffectual" to "4=very effectual." The data values represent the number of participants who indicated the intervention was "3 = Effective" or "4 = Very Effective."
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Participants are randomized to interventional arm which is seven-day intervention that requires them to download mobile app to complete educational courses each day. Participants are required to complete pre-and post-tests as part of the study. The intervention encourages education on mammogram needs.
  Educational mobile app: 7 day educational course to educate American Indian women to receive regular mammogram.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 60
Participants | 62 | 55
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .001, t-test, 2 sided — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Adverse events were not collected or reviewed for participants
Description: No adverse events were collected or reported on participants
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Research within a single tribe, like the Yankton Sioux Tribe, offers valuable insights into that community's unique dynamics. However, these findings cannot be broadly generalized. Each tribe has distinct traditions, languages, and community structures that shape health behaviors and outcomes, making cross-tribal generalization challenging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05530603/Prot_003.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT05530603/SAP_004.pdf
  • Informed Consent Form: Experimental Group (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT05530603/ICF_005.pdf
  • Informed Consent Form: Control Group (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT05530603/ICF_006.pdf